CLINICAL TRIAL: NCT04938414
Title: Inhibition of Caspase-1 Reduces Pyroptotic Neuroinflammation and Tissue Factor-Induced Cerebrospinal Fluid Circulation Impairment After Subarachnoid Hemorrhage
Brief Title: Investigate the Relationship Between Inflammatory and Coagulation in SAH CSF
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-892
Record Dates: First submitted 2021-06-21; First posted 2021-06-24 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-06

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: subarachnoid hemorrhage; coagulation; inflammation
MeSH Terms: conditions — Subarachnoid Hemorrhage; Thrombosis; Inflammation | interventions — Spinal Puncture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- subarachnoid hemorrhage: Patients with subarachnoid hemorrhage
  Interventions: Diagnostic Test: Lumbar puncture
- Control: patients with non-neurological diseases
  Interventions: Diagnostic Test: Lumbar puncture

INTERVENTIONS:
Diagnostic Test: Lumbar puncture — Lumbar puncture to obtain the cerebrospinal fluid and for diagnostic test

SUMMARY:
Investigate the role of inflammasome and blood coagulation response in human cerebrospinal fluid after subarachnoid hemorrhage.

DETAILED DESCRIPTION:
Investigate the role of inflammasome and blood coagulation response in human cerebrospinal fluid after subarachnoid hemorrhage (SAH).

1.40 patients with SAH will be included. The CSF will used for ELISA test for inflammatory factors and cogulation factors.

2.CSF obtained from 4 patients with non-neuroloogical disease with 4 addittional SAH patients will be used for Mass Spectrometry

ELIGIBILITY:
Inclusion Criteria:

* SAH patients with modified Fisher Scale 3-4.

Exclusion Criteria:

* Patients with history of CNS disease (e.g., stroke, traumatic brain injury, CNS infection) or accompanied by serious comorbidities before SAH onset (e.g., severe coagulation disorders, malignant tumor, uncontrollable heart disease, and hypertension) or other organ dysfunctions within 6 months were excluded from the study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with SAH
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | evaluated 1day after discharge
  Length of hospital stay
modified Rankin Scale | evaluated 1day after discharge
  modified Rankin Scale (mRS) at discharge. mRS ranging from 0-5, higher represents worse
Glasgow Outcome Scale | evaluated 1day after discharge
  Glasgow Outcome Scale (GOS) at discharge, GOS ranging from 0-5, higher represents better

CONTACTS AND LOCATIONS:
Overall Officials: Yuanjian Fang, M.D, Study Chair — Zhejiang Univerisity
Locations (1):
- Second affiliated hosipital of zhejiang univerisity school of medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No